CLINICAL TRIAL: NCT05807295
Title: The Effect of Relaxation Program on Coping With Stress and Anxiety Levels of Caregivers of Children With Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Çiğdem Sarı Öztürk, Gazi University, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1503
Record Dates: First submitted 2023-03-15; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Caregivers With a Child Followed up With a Cancer Diagnosis
MeSH Terms: interventions — Relaxation Therapy; Caregivers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): caregivers receiving a relaxation program
  Interventions: Other: Relaxation Program
- Control group (No Intervention): the group that did not receive any training

INTERVENTIONS:
Other: Relaxation Program — The relaxation program will include progressive muscle relaxation exercises and videos for relaxation. Videos will be sent to caregivers' social media accounts. Initial applications will be implemented with caregivers. The relaxation program is planned to last 6 weeks. The program is planned to last 8 weeks in total, with pre-test and post-test applications.
  Other Names: The relaxation program for caregivers
  Arms: Intervention

SUMMARY:
This research will be carried out to determine the effect of the relaxation program applied to the caregivers of children followed by the diagnosis of cancer on the levels of caregivers' anxiety and coping with stress. The research will be conducted in a single-blind parallel-group randomized controlled trial design. A relaxation program including progressive muscle relaxation exercises will be applied to caregivers. The application will be carried out by sending muscle relaxation videos and videos for relaxation to mothers. The relaxation program is planned to last approximately 6 weeks

DETAILED DESCRIPTION:
In this study, a relaxation program will be applied to mothers who have a child followed up with a cancer diagnosis. The relaxation program will include progressive muscle relaxation exercises and videos for relaxation. Initial applications will be implemented with caregivers. The relaxation program is planned to last 6 weeks. The program is planned to last 8 weeks in total, with pre-test and post-test applications. Caregivers will then be asked to perform the treatments each week. Coping with Stress and State-Trait Anxiety Scale will be used at the beginning and end of the program.

ELIGIBILITY:
Inclusion criteria

* The child has received cancer treatment for at least two months,
* Those who have internet access on their smartphone or computer
* Those who can continue the work for six weeks (doing progressive relaxation exercises at least 2 times a week)

Exclusion Criteria:

* Those whose children/caregivers are in the terminal period,
* Those whose child/caregiver has not received chemotherapy treatment,
* Those who take medication for anxiety or use one of the complementary medicine approaches.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-13 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
coping with stress | Change from Baseline level of Coping with stress to 8 weeks (change is being assessed)
  The scale is a 23-item self-report measure of anxiety using a 5-point Likert-type scale. The scale does not have a cut-off point. The higher the score obtained from the scale, the better the coping is determined.
Anxiety | Change from Baseline level of Spielberger State-Trait Anxiety to 8 weeks (change is being assessed)
  The scale is a 20-item self-report measure of anxiety using a 4-point Likert-type scale (from 0 to 3 points) for each item. The total score obtained from the scale varies between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozturk CS, Katikol E. Effect of mHealth-based relaxation program on stress coping and anxiety levels in mothers of children with cancer: A randomized controlled study. Patient Educ Couns. 2024 Jun;123:108247. doi: 10.1016/j.pec.2024.108247. Epub 2024 Mar 11. PMID 38471311